CLINICAL TRIAL: NCT07305285
Title: An Investigation Into the Effects and Mechanisms of Nursing Based on the Roy Adaptation Model on Psychological Status and Quality of Life in Patients Experiencing Facial Paralysis After Surgery for Giant Acoustic Neuroma
Brief Title: Roy Adaptation Model Improves Mood and QOL After Giant Acoustic Neuroma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WestChinaH-HX-2025-02
Record Dates: First submitted 2025-12-02; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Acoustic Neuroma; Facial Paralysis
Keywords: Roy Adaptation Model; Psychological state; Quality of life; Stress cytokines
MeSH Terms: conditions — Neuroma, Acoustic; Facial Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): RAM-Based Nursing + RAM Follow-Up Care：Core intervention (8 weeks): As described in the original protocol (four adaptation modes: physiological, self-concept, role function, interdependence).
  * Long-term follow-up (week 9 to 1 year):
  * Monthly online consultations (20-30 min/time): Via WeChat or video call to assess adaptation status (physical symptoms, psychological state, social participation); adjust self-management plans (e.g., facial muscle training intensity, psychological coping strategies).
  * Quarterly face-to-face visits (40-60 min/time): Conduct comprehensive assessment of facial nerve function (HB grade re-evaluation), psychological state, QoL, and electrophysiological function; organize peer support group meetings (semi-annually) to share long-term recovery experiences; strengthen family support guidance.
  Interventions: Behavioral: RAM-Based Nursing + RAM Follow-Up Care
- Control group (No Intervention): Routine Nursing + Routine Follow-Up
  * Core intervention (8 weeks): As described in the original protocol (postoperative basic care, standardized facial muscle training, health education, brief psychological support).
  * Long-term follow-up (week 9 to 1 year): Quarterly telephone follow-up (10-15 min/time) to inquire about facial function, psychological status, and adherence to training; provide verbal health education and guidance when necessary.

INTERVENTIONS:
Behavioral: RAM-Based Nursing + RAM Follow-Up Care — Core intervention (8 weeks): As described in the original protocol (four adaptation modes: physiological, self-concept, role function, interdependence).
  * Long-term follow-up (week 9 to 1 year):
  * Monthly online consultations (20-30 min/time): Via WeChat or video call to assess adaptation status (physical symptoms, psychological state, social participation); adjust self-management plans (e.g., facial muscle training intensity, psychological coping strategies).
  * Quarterly face-to-face visits (40-60 min/time): Conduct comprehensive assessment of facial nerve function (HB grade re-evaluation), psychological state, QoL, and electrophysiological function; organize peer support group meetings (semi-annually) to share long-term recovery experiences; strengthen family support guidance.
  Arms: Intervention Group

SUMMARY:
he goal of this randomized controlled trial is to learn if the Roy Adaptation Model (RAM) nursing program improves anxiety, depression, and quality of life in adults who have recently developed facial palsy. It will also learn about changes in stress-related blood markers. The main questions it aims to answer are: Does 12-week RAM nursing lower anxiety and depression scores compared with routine nursing? Does RAM nursing raise quality-of-life scores and beneficially alter serum levels of cortisol, IL-6, TNF-α, serotonin, and dopamine? Researchers will compare RAM nursing (one-to-one education, cognitive-behavioral support, facial-movement training, family counseling, and phone follow-up) to routine facial-palsy education only.

Participants will:

Receive either RAM nursing or routine nursing for 12 weeks Complete anxiety, depression, and quality-of-life questionnaires at baseline and week 12 Provide blood samples at baseline and week 12 to measure stress and inflammation markers

ELIGIBILITY:
Inclusion Criteria:

* Confirmed GAN by preoperative MRI (tumor diameter >4 cm) and postoperative pathological examination;
* Postoperative facial paralysis diagnosed by neurological examination, with House-Brackmann (HB) grade ≥Ⅱ;
* Age 18-65 years;
* Conscious, with normal cognitive function (Mini-Mental State Examination score ≥24), able to communicate and complete questionnaires independently;
* No history of psychological disorders or antidepressant/anxiolytic use before surgery;
* Signed informed consent.

Exclusion Criteria:

* Preoperative facial paralysis, facial nerve palsy, or other facial muscle diseases;
* History of schizophrenia, bipolar disorder, or other mental illnesses;
* Severe postoperative complications (e.g., intracranial infection, hemorrhage, cerebrospinal fluid leakage) requiring reoperation;
* Pregnancy or lactation;
* Severe liver, kidney, or cardiovascular diseases;
* Loss to follow-up or refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Self-Rating Anxiety Scale (SAS) | 1 year
  all are 20 items. The total score ranges from 20 to 80. A cut-off score of 50 indicates significant anxiety (scores ≥50 suggest anxiety symptoms). the higher the score, the worse the outcome
Self-Rating Depression Scale (SDS) | 1 year
  all are 20 items. The total score ranges from 20 to 80. A cut-off score of 53 indicates significant depression (scores ≥53 suggest depressive symptoms). the higher the score, the worse the outcome
World Health Organization Quality of Life-Brief(WHOQOL-BREF) | 1 year
  1. Reverse Scoring: For item 6 (pain/discomfort), reverse the score (1=5, 2=4, 3=3, 4=2, 5=1) because higher scores on this item indicate poorer quality of life. All other items are scored as per the original response.
  2. Domain Scores: Calculate the average score for each domain (Physical Health: Items 1-8; Psychological Health: Items 9-14; Social Relationships: Items 15-17; Environmental Domain: Items 18-26).
  3. Standardization: Convert each domain average score to a standard score (0-100) using the formula: Standard Score = [(Average Score - 1) / 4] × 100. Higher standard scores indicate better quality of life in that domain.

SECONDARY OUTCOMES:
Facial Nerve Electrophysiological Indicators | 1 year
  Assessed at baseline, 8 weeks, 6 months, and 1 year using a neuroelectromyography (EMG) instrument (Nicolet VikingSelect, USA) by a specialized neurologist blinded to group allocation:

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Protocol and Informed consent